CLINICAL TRIAL: NCT01772082
Title: Randomized Study of Use of Internet Mediated Walking Program and Pedometer in COPD
Brief Title: Use of Internet Mediated Walking Program and Pedometer in COPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Boston Healthcare System (U.S. Federal Agency)
Collaborators: University of Michigan (Other)
Responsible Party: Principal Investigator, Marilyn Moy, Associate Professor of Medicine, VA Boston Healthcare System
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ESCFull2328
Record Dates: First submitted 2013-01-16; First posted 2013-01-21 (Estimated); Last update posted 2017-03-14 (Actual); Status verified 2017-03

CONDITIONS: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pedometer alone (Active Comparator): pedometer
  Interventions: Behavioral: Internet mediated walking program
- Pedometer plus website (Experimental): pedometer and website
  Interventions: Behavioral: Internet mediated walking program

INTERVENTIONS:
Behavioral: Internet mediated walking program

SUMMARY:
Persons with COPD are randomized to pedometer versus pedometer plus Internet mediated website to promote walking and physical activity. Primary outcome is daily step counts. Intervention lasts 3 months.

ELIGIBILITY:
Inclusion Criteria:

COPD, ability to walk, has Internet access

Exclusion Criteria:

COPD exacerbation in previous 4 weeks

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2012-04-30 (Actual); Primary Completion 2016-01-06 (Actual); Study Completion 2017-02-02 (Actual)

PRIMARY OUTCOMES:
Daily Step Counts | pre and 3 months post
  measured by pedometer

CONTACTS AND LOCATIONS:
Locations (1):
- VABoston Healthcare System, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Berube MN, Robinson SA, Wan ES, Mongiardo MA, Finer EB, Moy ML. Physical Activity and Systemic Biomarkers in Persons With COPD: Insights from a Web-Based Pedometer-Mediated Intervention. Chronic Obstr Pulm Dis. 2024 Jul 25;11(4):369-381. doi: 10.15326/jcopdf.2023.0472. PMID 38809105
- [Derived] Robinson SA, Wan ES, Shimada SL, Richardson CR, Moy ML. Age and Attitudes Towards an Internet-Mediated, Pedometer-Based Physical Activity Intervention for Chronic Obstructive Pulmonary Disease: Secondary Analysis. JMIR Aging. 2020 Sep 9;3(2):e19527. doi: 10.2196/19527. PMID 32902390
- [Derived] Wan ES, Kantorowski A, Polak M, Kadri R, Richardson CR, Gagnon DR, Garshick E, Moy ML. Long-term effects of web-based pedometer-mediated intervention on COPD exacerbations. Respir Med. 2020 Feb;162:105878. doi: 10.1016/j.rmed.2020.105878. Epub 2020 Jan 11. PMID 32056676
- [Derived] Robinson SA, Shimada SL, Quigley KS, Moy ML. A web-based physical activity intervention benefits persons with low self-efficacy in COPD: results from a randomized controlled trial. J Behav Med. 2019 Dec;42(6):1082-1090. doi: 10.1007/s10865-019-00042-3. Epub 2019 Apr 12. PMID 30980223
- [Derived] Wan ES, Kantorowski A, Homsy D, Kadri R, Richardson CR, Mori D, Moy ML. Self-reported task-oriented physical activity: A comparison with objective daily step count in COPD. Respir Med. 2018 Jul;140:63-70. doi: 10.1016/j.rmed.2018.05.012. Epub 2018 May 19. PMID 29957283